CLINICAL TRIAL: NCT06900101
Title: Multimodal Monitoring Study in Neuro Critical Care
Acronym: MultiCU
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 713
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Subarachnoidal Hemorrhage; Intacranial Hypertension; Acute Trauma Brain Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Patients admitted in neurocritical care in Pierre Wertheimer hospital, following acute brain injury,
  Interventions: Other: Study the evolution and correlation between cerebral autoregulation index

INTERVENTIONS:
Other: Study the evolution and correlation between cerebral autoregulation index — Objective n°1: Study the correlation between autoregulation index:
  The investigators will look for a correlation between several auroregulation index such as the PRx, ORx and Cox.
  Objective n°2: Evaluation and detection of EEG prognostic patterns: The investigators will look for quantitaive EEG changes during the early phase of acute brain injuries.

SUMMARY:
During the first week after an acute cerebral injury, neurologic clinical exam is often irrelevant, limited by sedation use or spontaneous consciousness disorders.

Hence, neurological monitoring of brain oxygen consumption, metabolic disorders, electrical activity is used to follow and prevent delayed cerebral injuries. Among those instruments, numerous are often described: intra cranial pressure monitoring, brain tissue oxygen pressure monitoring, scalp electroencephalography, continuous electroencephalography and Near infrared Red Spectroscopy (NIRS).

Even if the value of some of those technologies are well known, many remain part of a research domain. Here we will not only try to study the correlation between different cerebral autoregulation's index described in the scientific literature but also will we try to identify and describe EEG and cardiorespiratory changes during the first week following brain injury. The objective of this study is to investigate the pathophysiology of acute brain injury and explore potent biomarkers of multimodal monitoring during the first week following acute brain injury.

ELIGIBILITY:
Inclusion Criteria:

* - Patients hospitalized in neurologic critical care in Wertheimer Hospital, Bron
* Monitored with the CNS MOBERG® monitoring system

Exclusion Criteria:

* - Refusal to participate
* Patients under legal protection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in neuro critical care, in Pierre Wertheimer hospital, for acute brain injury and monitored by MOBERG® system.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between ORx and PRx | Multimodal neuro monitoring is used from 1 to 15 days after the acute brain injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pierre Wertheimer, France, Bron, France